CLINICAL TRIAL: NCT04668495
Title: Impact of Timing of Pharmacodynamic Assessments on Measures of Platelet Reactivity in Patients Undergoing Percutaneous Coronary Intervention Treated With Cangrelor
Brief Title: Impact of Timing of PD Assessments on Measures of Platelet Reactivity in Patients Undergoing PCI Treated With Cangrelor
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: Cangrelor Timing
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cangrelor Group: This is the study cohort that the blood sample will be obtained from. There are no interventions

SUMMARY:
This study is assessing the impact of timing of PD assessments on measures of platelet reactivity in patients undergoing PCI treated with cangrelor.

DETAILED DESCRIPTION:
Cangrelor is characterized by reversible binding to the P2Y12 receptor and is promptly inactivated through dephosphorylation by ectonucleotidase leading to its very short plasma half-life. Consequently the timing at which PD assessments are performed after blood sample collection may impact measures of platelet reactivity in patients treated with cangrelor. We therefore hypothesize that measures of platelet inhibitory effects observed in cangrelor treated patients will reduce with time following blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* CAD patients (stable CAD, NSTE-ACS, or STEMI) undergoing PCI and treated with cangrelor per standard of care.
* Treated with aspirin prior to the PCI procedure per standard of care

Exclusion Criteria:

* Treatment with an oral P2Y12 inhibitor (clopidogrel, prasugrel or ticagrelor) within past 10 days
* Treatment with oral anticoagulation (vitamin K antagonist, dabigatran, apixaban, rivaroxiban) within past 3 days
* Treatment with a glycoprotein IIb/IIIa inhibitor during PCI
* Fibrinolytics within 48 hours
* Known hemoglobin<10 gm/dL
* Known platelet count <80x106/mL
* Active bleeding or hemodynamic instability
* Known end stage renal disease on hemodialysis
* Known severe hepatic dysfunction

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing percutaneous coronary intervention (PCI) and have been treated with cangrelor per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Change in platelet reactivity | wiithin 30 min, 1 hour, 2 hours, and 4 hours of blood sampling
  measure of change platelet reactivity at time points

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, MD, PhD, Principal Investigator — Professor of Medicine
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franchi F, Rollini F, Galli M, Been L, Ghanem G, Shalhoub A, Rivas A, Zhou X, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Bass TA, Angiolillo DJ. Impact of Timing of Pharmacodynamic Assessment on Platelet Reactivity in Patients Treated With Cangrelor. JACC Cardiovasc Interv. 2021 Nov 8;14(21):2410-2412. doi: 10.1016/j.jcin.2021.07.051. No abstract available. PMID 34736741